CLINICAL TRIAL: NCT05793242
Title: Immediate and 24-hour Effects of the HyperVolt Device, Body Tempering, and Cupping Compared to Static Stretching of the Hamstring Muscles to Increase Lower Extremity Range of Motion
Brief Title: Immediate and 24-hour Effects of HyperVolt, Body Tempering, and Cupping Compared to Stretching on Hamstring Flexibility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Cathy Arnot, Project Director, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00125174
Record Dates: First submitted 2023-03-15; First posted 2023-03-31 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Hamstring Contractures; Muscle Tightness
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Static stretching (Active Comparator): The static stretch group participants will perform a self-facilitated stretch by looping a strap around the heel of their foot and grasping it with both hands followed by pulling the strap to raise the fully extended leg into hip flexion. The participant will then lift the leg until they reach their maximal tolerable point and then alternate between periods of resting and stretching for a total of 5 minutes.
  Interventions: Other: Static stretching
- Hypervolt (Experimental): The HyperVolt percussive massage group participants will receive a therapist-performed HyperVolt technique to the hamstrings for a period of 5 minutes.
  Interventions: Device: Hypervolt
- Body tempering (Experimental): The body tempering group participants will receive a therapist-performed body tempering technique to the hamstrings for a period of 5 minutes.
  Interventions: Device: Body Tempering
- Dry cupping (Experimental): The dry cupping group participants will receive a therapist-performed dry cupping technique to the hamstrings for a period of 5 minutes.
  Interventions: Device: Dry cupping

INTERVENTIONS:
Device: Hypervolt — HyperVolt Percussive Massage Device: this will be performed by a physical therapist while the participant is prone. The physical therapist will apply a vibrating device to the back of the thigh with moderate pressure while continuously moving the device for 5 minutes.
  Arms: Hypervolt
Device: Body Tempering — Body Tempering:this will be performed by a physical therapist while the participant is prone. The physical therapist will apply a moderately heavy metal device to the back of the thigh while continuously moving the device for 5 minutes.
  Arms: Body tempering
Device: Dry cupping — Dry Cupping: This will be performed by a physical therapist while the participant is prone. The physical therapist will apply several negative pressure devices to the back of your thigh for 5 minutes.
  Arms: Dry cupping
Other: Static stretching — Participants will perform a static stretch on their lower extremity. This stretch will be performed by having the participant loop a strap around their heel and grasping it with both hands followed by pulling the strap to raise the fully extended leg into hip flexion. The participant will be instructed to lift the leg until they reach their maximal tolerable point and then to hold the position for 30 seconds. They will then lower the extremity to the table and rest for 15 seconds This self-stretch sequence will be performed for 7 cycles so that the total intervention was equal to the intervention time of the other group (5 minutes).7
  Arms: Static stretching

SUMMARY:
The purpose of this study is to compare the effects of the HyperVolt percussive massage device, body tempering, and dry cupping to static stretching of the hamstrings of healthy adults aged 18-39 years on the active knee extension and back saver sit-and-reach test.While these modalities are frequently used in healthcare settings there is a paucity of research regarding effectiveness. If the effects on flexibility are comparable, patients could save time and money by performing static stretching.

DETAILED DESCRIPTION:
Our study aims to compare the effects of the HyperVolt percussive massage device (HyperVolt), body tempering, and dry cupping compared to static stretching on flexibility and range of motion (ROM), specifically in those with active hamstring ROM limitations. Those individuals from the University of South Carolina community who are interested in becoming study participants will be identified by means of announcements made in the Seminar in Physical Therapy course which is attended by all Physical Therapy students, faculty, and staff each week. Interested individuals will be provided with Dr.Cathy Arnot's email address in order to schedule an evaluation session to determine whether or not they meet the study's inclusion and exclusion criteria. A flyer will also be posted in the Blatt PE Building with Sean Edmonds' contact information included. Interested individuals that contact Sean will be scheduled for screening by Dr.Cathy Arnot. Participants will be assigned to either the HyperVolt percussive massage device (HyperVolt) group, body tempering group, dry cupping group, or static stretching group via blocked randomization for sex and age, with at least twenty participants being placed into each group. The HyperVolt percussive massage group participants will receive a therapist-performed HyperVolt technique for a period of 5 minutes. The body tempering group participants will receive a therapist-performed body tempering technique for a period of 5 minutes. The dry cupping group participants will receive a therapist-performed dry cupping technique for a period of 5 minutes. The static stretch group participants will perform a self-facilitated stretch by looping a strap around the heel of their foot and grasping it with both hands followed by pulling the strap to raise the fully extended leg into hip flexion. The participant will then lift the leg until they reach their maximal tolerable point and then alternate between periods of resting and stretching for a total of 5 minutes. Measurements will be assessed at three time points: Immediately before the intervention, immediately after the intervention, and 24 hours after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Shortened hamstring length
* Male participants will display ≤141 degrees of knee extension
* Female participants will display ≤152 degrees of knee extension

Exclusion Criteria:

* history of knee injury
* hypertension
* thrombophlebitis
* inflammation
* myositis ossificans
* osteomyelitis
* open wounds
* unhealed fractures
* hematoma or hemophilia
* pregnancy
* cancer
* burns or skin grafts
* varicose veins
* synovitis
* currently taking any anticoagulation medications
* rheumatoid arthritis
* osteoporosis
* any other condition that would prevent safe participation

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Active Knee Extension Test (AKE) | Immediately after intervention
  The Active Knee Extension (AKE) Test measures will be conducted by a pair of graders that will be blinded to the intervention applied to the study participants. Participants will have an axis of rotation labeled at the lateral aspect of the knee joint midline. The participant will be instructed to lie down on the table in the supine position. One of the test graders will assist the participant in performing and maintaining 90-degrees of hip flexion throughout this test. The participant will be instructed to extend at the knee as much as possible and told to hold the position for the second grader to measure the knee extension ROM using a goniometer. A total of 3 measurements will be conducted, with the last 2 recorded for data analysis.
Active Knee Extension Test (AKE) | 24 hours after the intervention
  The Active Knee Extension (AKE) Test measures will be conducted by a pair of graders that will be blinded to the intervention applied to the study participants. Participants will have an axis of rotation labeled at the lateral aspect of the knee joint midline. The participant will be instructed to lie down on the table in the supine position. One of the test graders will assist the participant in performing and maintaining 90-degrees of hip flexion throughout this test. The participant will be instructed to extend at the knee as much as possible and told to hold the position for the second grader to measure the knee extension ROM using a goniometer. A total of 3 measurements will be conducted, with the last 2 recorded for data analysis.
Back-Saver Sit-and-Reach Test | Immediately after intervention
  The Back-Saver Sit-and-ReachTest will be conducted by a pair of graders that will be blinded to the intervention group of the study participants. A box will be utilized with a ruler placed on top of the box with 9 inches protruding out towards the participant. The ruler will run parallel to the direction of forward movement by the participant. When instructed, the tested lower extremity will remain fully extended at the knee with the plantar side of the foot flat up against the wall of the box. The contralateral non-tested leg will be flexed at the knee, resulting in the plantar side of the foot flat down against the floor. The foot of the non-tested leg will be placed within 2 to 3 inches away from the fully extended tested leg and remain planted at all times during testing procedures. Participants will be instructed to reach forward as far as possible with arms fully extended, back straight, and head up.
Back-Saver Sit-and-Reach Test | 24 hours after the intervention
  The Back-Saver Sit-and-ReachTest will be conducted by a pair of graders that will be blinded to the intervention group of the study participants. A box will be utilized with a ruler placed on top of the box with 9 inches protruding out towards the participant. The ruler will run parallel to the direction of forward movement by the participant. When instructed, the tested lower extremity will remain fully extended at the knee with the plantar side of the foot flat up against the wall of the box. The contralateral non-tested leg will be flexed at the knee, resulting in the plantar side of the foot flat down against the floor. The foot of the non-tested leg will be placed within 2 to 3 inches away from the fully extended tested leg and remain planted at all times during testing procedures. Participants will be instructed to reach forward as far as possible with arms fully extended, back straight, and head up.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy F Arnot, DPT, Study Director — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blazevich AJ, Gill ND, Kvorning T, Kay AD, Goh AG, Hilton B, Drinkwater EJ, Behm DG. No Effect of Muscle Stretching within a Full, Dynamic Warm-up on Athletic Performance. Med Sci Sports Exerc. 2018 Jun;50(6):1258-1266. doi: 10.1249/MSS.0000000000001539. PMID 29300214
- [Result] Aguilar AJ, DiStefano LJ, Brown CN, Herman DC, Guskiewicz KM, Padua DA. A dynamic warm-up model increases quadriceps strength and hamstring flexibility. J Strength Cond Res. 2012 Apr;26(4):1130-41. doi: 10.1519/JSC.0b013e31822e58b6. PMID 22446678
- [Result] Konrad A, Glashuttner C, Reiner MM, Bernsteiner D, Tilp M. The Acute Effects of a Percussive Massage Treatment with a Hypervolt Device on Plantar Flexor Muscles' Range of Motion and Performance. J Sports Sci Med. 2020 Nov 19;19(4):690-694. eCollection 2020 Dec. PMID 33239942
- [Result] Taber CB, Colter RJ, Davis JJ, Seweje PA, Wilson DP, Foster JZ, Merrigan JJ. The Effects of Body Tempering on Force Production, Flexibility and Muscle Soreness in Collegiate Football Athletes. J Funct Morphol Kinesiol. 2022 Jan 11;7(1):9. doi: 10.3390/jfmk7010009. PMID 35076554
- [Result] Williams JG, Gard HI, Gregory JM, Gibson A, Austin J. The Effects of Cupping on Hamstring Flexibility in College Soccer Players. J Sport Rehabil. 2019 May 1;28(4):350-353. doi: 10.1123/jsr.2017-0199. Epub 2018 Dec 4. PMID 29364033
- [Result] Gunn LJ, Stewart JC, Morgan B, Metts ST, Magnuson JM, Iglowski NJ, Fritz SL, Arnot C. Instrument-assisted soft tissue mobilization and proprioceptive neuromuscular facilitation techniques improve hamstring flexibility better than static stretching alone: a randomized clinical trial. J Man Manip Ther. 2019 Feb;27(1):15-23. doi: 10.1080/10669817.2018.1475693. Epub 2018 Aug 1. PMID 30692839